CLINICAL TRIAL: NCT02594423
Title: Management of Active and Established Corneal Neovascularisation to Prevent Visual Impairment
Brief Title: Strategies for Management of Corneal Neovascularisation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15070; 2015-003180-11 (EudraCT Number)
Record Dates: First submitted 2015-10-27; First posted 2015-11-03 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Corneal Neovascularisation
MeSH Terms: conditions — Corneal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fine needle Diathermy (Active Comparator): Fine needle Diathermy(FND) will be applied under topical anaesthesia under an operating microscope. This involves the insertion of a fine corneal suture needle in the vicinity of the vessels and using this as an extension of the probe of a monopolar cautery to deliver the energy in the corneal tissue at the site at which it is required to occlude the vessels.
  Interventions: Device: Fine Needle Diathermy
- Fine Needle Diathermy and Bevacizumab (Active Comparator): Fine needle Diathermy(FND) will be applied under topical anaesthesia under an operating microscope. This involves the insertion of a fine corneal suture needle in the vicinity of the vessels and using this as an extension of the probe of a monopolar cautery to deliver the energy in the corneal tissue at the site at which it is required to occlude the vessels. Patients will receive subconjunctival injections of bevacizumab in the conjunctiva near the limbus in the quadrant(s) affected (total volume of between 0.2 ml-0.3 ml of the 2.5 mg/0.1 ml solution). The subconjunctival injections will be administered after FND in the same treated quadrants.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Device: Fine Needle Diathermy — Fine needle diathermy is a surgical procedure that is used in the treatment of corneal NV. It is a safe and effective method for corneal vessels occlusion.
  Arms: Fine needle Diathermy
Drug: Bevacizumab — Bevacizumab is a humanized monoclonal antibody that binds to isoforms of VEGF-A .
  Other Names: Avastin(BEVACIZUMAB)
  Arms: Fine Needle Diathermy and Bevacizumab

SUMMARY:
The cornea is the transparent window of the eye, which allows light to enter into the eye and also contributes to the focusing of the light rays. One of the major factors responsible for its transparency is the lack of blood vessels. However, following inflammation new blood vessels (corneal vascularisation [CVas]) grow into the cornea affecting its transparency and impairing vision. CVas leads to further damage in the form of scarring,oedema,fat deposition and is a major cause of corneal graft rejection.

In 2000 with ethical approval (OY129801) the investigators developed and published a clinical technique called Fine Needle Diathermy occlusion of corneal vessels (FND). This has proven very successful for occluding established vessels and is practiced in many centers across the world. Recently it has been demonstrated that by inhibiting a chemical stimulant of vessel formation called vascular endothelial growth factor(VEGF) active new vessel growth in the retina can be suppressed. The approach is also being used for corneal new vessels. Bevacizumab (Avastin) is a chemical inhibitor of VEGF and is used extensively to treat retinal new vessels in macular degeneration. Avastin has been shown to be effective and safe in treating corneal new vessels. The investigators propose to evaluate the efficacy and safety of FND alone and FND combined with Avastin in treatment of CVas.

DETAILED DESCRIPTION:
Corneal neovascularisation is a very common problem affecting both sexes at all ages and induced by differing underlying causes. It is considered to be the single most important risk factor for graft rejection. The process of angiogenesis, i.e. the formation of new blood vessels, is similar in any part of the body. Hence principles adopted to alleviate new blood vessels in one area can be applied to blood vessels in other areas using similar drugs.

Over the past 8 years a component necessary for angiogenesis, i.e Vascular endothelial growth factor (VEGF) has been targeted to induce regression of blood vessels in patients with cancer with an intravenous dosage of an anti-VEGF.

More recently, anti-VEGF therapies have targeted eye related neovascularisation, especially in the treatment of age related macular degeneration. This role has been expanded to include all other structures in the eye affected by angiogenesis such as neovascular glaucoma(Iris) and diabetic retinopathy(Retina).

Over the past few years attention has been drawn to the use of antiVEGF therapies to the surface of the eye. Many reports in international peer reviewed literature have commented on the use of anti VEGF therapy in the form of drops or injections on the surface of the eye, subconjunctivally and within the cornea. They have found drops and injections are safe, although injections appear to act more favourably. Avastin has been investigated for treating corneal new vessels and was proved to be both safe and effective.

Fine needle diathermy (FND) is a routine method for occluding corneal vessels that was developed in our department in 2000 and is used worldwide. It has been established that this technique is suitable for active and mature vessels.

However, the consequent transient tissue injury and inflammation can trigger further new vessel formation. Avastin is effective in occlusion of the active vessels only.It does not affect the established mature vessels. Hence if FND is combined with Avastin it is expected and hypothesized that a more efficient and lasting occlusion of vessels will be obtained. In this study, the investigators aim to investigate the combined action of Avastin and fine needle diathermy in occlusion of corneal vessels. The actual incidence of corneal neovascularisation in the UK is unknown but American studies suggest up to 1.4 million people are affected with sight threatening complications on annual basis. These blood vessels arise from a multitude of causes, including viral infections, corneal injuries, chronic inflammation and as a result of corneal transplantation. Conventional therapies at the present time include surgical occlusion of the blood vessels with a diathermy or laser or chronic use of steroids. The latter option is a associated with potential sight threatening complications such as glaucoma.

This study will generate data to inform further controlled studies towards establishing Avastin and fine needle diathermy as the treatment of choice for corneal new vessels.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Able to give informed consent
* With corneal neovascularisation non responsive or not suitable for conventional steroid therapy
* Use of effective contraception in females of childbearing age

Exclusion Criteria:

* Patients under 18 years of age
* Patients unable or refusing to provide informed consent
* Patients who are needle phobic
* Pregnant women, women aiming for conception and breastfeeding women
* Patients with hypersensitivity to the active substance or to any of the excipients
* Patients with active or suspected ocular or periocular infections.
* Patients with active severe intraocular inflammation.
* Patients with raised intraocular pressure or on glaucoma medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Decreased corneal neovascularisation | 6 months
  A comparison of total vascularisation of the corneal area as measured by our grading system (Faraj LA et al, 2015) before and after treatment.

SECONDARY OUTCOMES:
Improved/maintained Snellen's visual acuity | 10 months
  Visual acuity is assessed using Snellen chart and vision is expressed in LOGMAR units
Decreased corneal opacity related to lipid deposition | 10 months
  The response to treatment will be judged clinically by biomicroscopy examination and quantitatively by comparison with pre-treatment slit lamp photographs. The comparison of the pre and post treatment slit lamp images will be done by two independent blind reviewers.
Reduced episodes of graft rejection(in corneal graft patients) | 10 months
  Number of rejection episodes will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Harminder S Dua, Professor, Principal Investigator — University of Nottingham